CLINICAL TRIAL: NCT01997307
Title: Age at Menopause and Severity of Coronary Artery Disease Among Postmenopausal Women With Acute Coronary Syndromes
Brief Title: The LADIES Acute Coronary Syndromes Study
Acronym: Ladies ACS
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 117/2013
Record Dates: First submitted 2013-09-14; First posted 2013-11-28 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2015-12

CONDITIONS: Acute Coronary Syndromes; Menopause
Keywords: acute coronary syndrome, coronary arteriography, menopause
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Stratification by gender and age, including 4 age categories: >=55-64 years
- Age >=65 to 74
- Age >=75 to 84
- Age >=85

SUMMARY:
The Ladies ACS study will investigate the relation between age at menopause and severity of coronary artery disease in menopausal women with acute coronary syndromes and clinical indication to coronary angiography.

DETAILED DESCRIPTION:
Multicenter prospective study in consecutive patients hospitalized with a wide spectrum of ACS and clinical indication to coronary angiography.

Consecutive patients older than 55 years with an ACS undergoing coronary angiography are eligible for the study, irrespective of subsequent revascularization. Eligible are women and men with a 2:1 enrolment ratio.

Patients will be stratified according to gender and age, including four age categories: 55-64, 65-74, 75-85 and >85 years. Each age category will include 200 patients, and enrolment in each category will be stopped once this number has been reached.

A specific electronic web-based CRF will collect clinical and procedural data. Clinical data input will take place at the participating Centers. Angiographic data input will be performed at rthe angiographic corelab, blinded of clinical data.

The e-CRF will collect data on

* the characteristics of the ACS
* the relevant risk factors for CAD and known prognostically relevant variables
* prior clinical history (prior MI, PCI, CABG, heart failure, stroke)
* in women fertility history will be captured by specific items, including age at first and last menstrual period, past use of oral contraceptives, ongoing and past hormone replacement therapy (HRT) and whether they had undergone a hysterectomy and/or oophorectomy, as well as information on the number of full-term pregnancies (the sum of live births and stillbirths). Age at menarche is defined as the age at the first menstrual period. Reproductive life span is automatically calculated calculated by subtracting the age at menarche from the age at menopause. The presence of hot flushes, their severity and duration in years will be also captured.

The extent of coronary artery disease will be evaluated at a central corelab using the Gensini score and the SYNTAX score

ELIGIBILITY:
Inclusion Criteria:

Patients >55 years of age with all of the following characteristics:

* symptoms suggestive of acute myocardial ischemia within the previous 48 hours.
* The diagnosis of an ACS must be confirmed by a typical rise and fall in serum troponin levels as defined by the Third Universal Definition of Myocardial Infarction.
* ECG signs of myocardial ischemia defined as either transient or persistent ST segment elevation or depression >0.5 mm (but >1 mm in the case of ST-segment elevation), or persistent and definite T-wave inversion >1 mm, including the pseudonormalization of a previously negative T-wave, in ≥2 contiguous leads.

Exclusion Criteria:

* none

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients older than 55 years with an acute coronary syndromes, undergoing coronary angiography are eligible for the study, irrespective of subsequent revascularization. Eligible are women and men with a 2:1 enrolment ratio.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Extent of coronary artery disease at angio corelab (Gensini and SYNTAX score) | 1 day
  The primary study end-point will be the severity of coronary artery disease, as appraised by the Gensini score

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Savonitto, MD, Study Chair — Division of Cardiology, Manzoni Hospital, Lecco; Giovanni Tortorella, MD, Principal Investigator — Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
Locations (1):
- Arcispedale Santa Maria Nuova- IRCCS, Reggio Emilia, Italy, Italy

REFERENCES:
- [Derived] Savonitto S, Morici N, Franco N, Misuraca L, Lenatti L, Ferri LA, Lo Jacono E, Leuzzi C, Corrada E, Aranzulla TC, Cagnacci A, Colombo D, La Vecchia C, Prati F; LADIES ACS Investigators. Age at menopause, extent of coronary artery disease and outcome among postmenopausal women with acute coronary syndromes. Int J Cardiol. 2018 May 15;259:8-13. doi: 10.1016/j.ijcard.2018.02.065. Epub 2018 Feb 21. PMID 29486998
- [Derived] Savonitto S, Colombo D, Franco N, Misuraca L, Lenatti L, Romano IJ, Morici N, Lo Jacono E, Leuzzi C, Corrada E, Aranzulla TC, Petronio AS, Bellia G, Romagnoli E, Cagnacci A, Zoccai GB, Prati F; LADIES ACS Study Investigators. Age at Menopause and Extent of Coronary Artery Disease Among Postmenopausal Women with Acute Coronary Syndromes. Am J Med. 2016 Nov;129(11):1205-1212. doi: 10.1016/j.amjmed.2016.05.031. Epub 2016 Jun 16. PMID 27321972